CLINICAL TRIAL: NCT02255760
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of MEDI3902 in Healthy Adults
Brief Title: Phase 1 Randomized Double-blind Placebo Controlled Study to Evaluate Safety and PK of MEDI3902 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5470C00002
Record Dates: First submitted 2014-09-16; First posted 2014-10-03 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: MEDI3902 for Prevention of P. Aeruginosa Pneumonia
Keywords: MEDI3902; Safety,; Pharmacokinetics,; Healthy Volunteers
MeSH Terms: interventions — gremubamab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MEDI3902 - Dose 1 (Experimental): Participants will receive a single intravenous (IV) dose of MEDI3902 infused for a minimum of 13 minutes on Day 1.
  Interventions: Drug: MEDI3902 - Dose 1
- MEDI3902 - Dose 2 (Experimental): Participants will receive a single IV dose of MEDI3902 infused for a minimum of 38 minutes on Day 1.
  Interventions: Drug: MEDI3902 - Dose 2
- MEDI3902 - Dose 3 (Experimental): Participants will receive a single IV dose of MEDI3902 infused for a minimum of 75 minutes on Day 1.
  Interventions: Drug: MEDI3902 - Dose 3
- MEDI3902 - Dose 4 (Experimental): Participants will received a single IV dose of MEDI3902 infused for a minimum of 150 minutes on Day 1.
  Interventions: Drug: MEDI3902 - Dose 4
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo by IV infusion up to a maximum of 12 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI3902 - Dose 1 — Participants will receive a single IV dose of MEDI3902 infused for a minimum of 13 minutes on Day 1.
  Other Names: MEDI3902
  Arms: MEDI3902 - Dose 1
Drug: MEDI3902 - Dose 2 — Participants will receive a single IV dose of MEDI3902 infused for a minimum of 38 minutes on Day 1.
  Other Names: MEDI3902
  Arms: MEDI3902 - Dose 2
Drug: MEDI3902 - Dose 3 — Participants will receive a single IV dose of MEDI3902 infused for a minimum of 75 minutes on Day 1.
  Other Names: MEDI3902
  Arms: MEDI3902 - Dose 3
Drug: MEDI3902 - Dose 4 — Participants will received a single IV dose of MEDI3902 infused for a minimum of 150 minutes on Day 1.
  Other Names: MEDI3902
  Arms: MEDI3902 - Dose 4
Other: Placebo — Participants will receive a single dose of placebo by IV infusion up to a maximum of 12 hours.
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, dose escalation study evaluating the safety and tolerability of a single ascending IV dose of MEDI3902 in healthy adult subjects 18 to 60 years of age.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, dose escalation study evaluating the safety and tolerability of a single ascending IV dose of MEDI3902 in healthy adult subjects 18 to 60 years of age. Approximately 40 subjects will be enrolled across 4 fixed dose cohorts at 1 study site. This study will last approximately 90 days, constituting a screening period of up to 28 days, 1 day of investigational product administration, and a 60 day safety follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 60 years at the time of screening
2. Written informed consent
3. Weight greater than or equal to (>=) 45 kilogram (kg) and less than or equal to (<=) 110 kg at screening
4. Healthy by medical history, physical examination, and baseline safety laboratory studies
5. Systolic blood pressure (BP) less than (<) 140 millimeter of mercury (mmHg) and diastolic BP < 90 mmHg at screening
6. Electrocardiogram (ECG) without clinically significant abnormalities at screening
7. Able to complete the follow-up period through Day 61 as required by the protocol.
8. Females of childbearing potential who are sexually active with a nonsterilized male partner must have used a highly effective method of contraception for at least 28 days prior to dosing with investigational product and must agree to continue using such precautions through Day 61 of the study.

Exclusion Criteria:

1. Acute (time-limited) illness, including fever 99.5 degree Fahrenheit (0^F), on day prior to or day of planned dosing
2. Any drug therapy within 7 days prior to Day 1 (except contraceptives or a single use of acetaminophen, aspirin, antihistamine, or combination over-the-counter (OTC) product that contains acetaminophen with an antihistamine, or OTC non-steroidal anti inflammatory agent at a dose equal to or lower than that recommended on the package). Vitamins and other nutritional supplements that are not newly introduced, ie, have been taken for at least 30 days prior to enrolment, are not exclusionary
3. Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 2 months prior to screening
4. Receipt of immunoglobulin or blood products within 6 months prior to screening
5. Receipt of any investigational product in the preceding 90 days or expected receipt of investigational product during the period of study follow-up, or concurrent participation in another interventional study Receipt of any vaccine within 7 days prior to investigational product dosing or planned receipt within 61 days after investigational product dosing except for influenza vaccine administered at least 28 days after dosing
6. Previous receipt of a mAb
7. Immunodeficiency due to illness, including human immunodeficiency virus (HIV) infection, or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening. HIV testing must be negative at screening
8. History of allergic disease or reactions likely to be exacerbated by any component of the investigational product
9. Either history of active infection with hepatitis B or C
10. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or serum creatinine above the upper limit of normal (ULN) or hemoglobin, white blood cell count, or platelet count below the lower limit of normal at screening and in the predose blood sample
11. Pregnant or nursing mother

13. History of alcohol or drug abuse within the past 2 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2015-04-20 (Actual); Study Completion 2015-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan S. Jafri, M.D., Study Director — MedImmune LLC; Martha Hernandez-Illas, MD, Principal Investigator — MRA Clinical Research, LLC
Locations (1):
- Research Site, South Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 131 participants were screened, of which 75 did not meet eligibility criteria and were considered as screen failures; and the remaining 56 participants were randomized into the study.
Groups:
- Placebo: Participants received a single dose of placebo by intravenous (IV) infusion up to a maximum of 12 hours.
- MEDI3902 - Dose 1: Participants received a single IV dose of MEDI3902 infused for a minimum of 13 minutes on Day 1.
- MEDI3902 - Dose 2: Participants received a single IV dose of MEDI3902 infused for a minimum of 38 minutes on Day 1.
- MEDI3902 - Dose 3: Participants received a single IV dose of MEDI3902 infused for a minimum of 75 minutes on Day 1.
- MEDI3902 - Dose 4: Participants received a single IV dose of MEDI3902 infused for a minimum of 150 minutes on Day 1.
Period: Overall Study
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Started | 14 | 3 | 15 | 15 | 9
Completed | 14 | 2 | 15 | 15 | 9
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who had received any dose of study drug were included in the as-treated population and subjects were analyzed according to the treatment they actually received.
Groups:
- Placebo: Participants received a single dose of placebo by IV infusion up to a maximum of 12 hours.
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4 | Total
Number analyzed (Participants) | 14 | 3 | 15 | 15 | 9 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (10.9) | 34.0 (9.5) | 40.9 (11.8) | 40.3 (12.4) | 39.8 (13.1) | 40.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 9 | 9 | 6 | 36
  Male | 5 | 0 | 6 | 6 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A TEAE is defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 to Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 14 | 3 | 15 | 15 | 9
Participants | 4 | 2 | 6 | 8 | 6

2. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment Emergent Adverse Events of Special Interest (TEAESIs)
Description: An AE is any untoward medical occurrence attributed to study drug in a participant who received investigational product. TESAE was an event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly that occurred after the initial receipt of the study drug. An AESI was one of scientific and medical interest specific to understanding of study product and may have required close monitoring and rapid communication by investigator to the sponsor. TEAESIs were collected from the time of dosing through Day 61 after the last dose of study drug and included anaphylaxis, other serious allergic reactions, infusion-related reactions, hepatic function abnormalities and immune complex disease.
Time Frame: Day 1 to Day 61
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 14 | 3 | 15 | 15 | 9
Participants
  TESAEs | 0 | 0 | 0 | 0 | 0
  TEAESIs | 0 | 0 | 4 | 6 | 5

3. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Any medically significant change in laboratory evaluations were recorded as adverse events. Following parameters were analyzed for laboratory examination: Hematology, serum chemistry, liver function, serum electrolytes and urinalysis.
Time Frame: Day 1 to Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 14 | 3 | 15 | 15 | 9
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital signs measurements included temperature, blood pressure (systolic and diastolic), pulse rate and respiratory rate.
Time Frame: Day 1 to Day 7
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 14 | 3 | 15 | 15 | 9
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Area Under the Serum Concentration-time Curve From Zero to Infinity (AUC [0-infinity])
Description: Area under the serum concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - infinity). The PK parameter AUC (0-inf) was estimated based on the serum concentrations of MEDI3902. Non-compartmental PK data analysis was performed to estimate the serum PK parameters of MEDI3902.
Time Frame: Pre-dose (24 hours prior to dose); at the end of the infusion, and 8 hours post infusion, and Days 2, 3, 7, 15, 22, 29, 43, and 61 post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: micrograms*day/milliliters
Arm/Group | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 3 | 15 | 15 | 8
micrograms*day/milliliters | 694 (133) | 2149 (625) | 4246 (1117) | 6540 (1817)

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for MEDI3902 After First Dose
Description: The PK parameter Cmax was estimated based on the serum concentrations of MEDI3902. Non-compartmental PK data analysis was performed to estimate the serum PK parameters of MEDI3902.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 3 | 15 | 15 | 8
micrograms/milliliter | 100 (6) | 207 (36) | 468 (134) | 838 (181)

7. Secondary Outcome: Terminal Phase Elimination Half-life (t1/2)
Description: The t1/2 is the time measured for the serum drug concentration of MEDI3902 to decrease by one half. The PK parameter t1/2 was estimated based on the serum concentrations of MEDI3902. Non-compartmental PK data analysis was performed to estimate the serum PK parameters of MEDI3902.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 3 | 15 | 15 | 8
Days | 7.2 (0.9) | 9.0 (2.1) | 9.4 (1.6) | 8.4 (0.8)

8. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug uniformly distributed to produce the desired serum concentration of a drug. The PK parameter Vss was estimated based on the serum concentrations of MEDI3902. Non-compartmental PK data analysis was performed to estimate the serum PK parameters of MEDI3902.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 3 | 15 | 15 | 8
milliliters | 3412 (107) | 4022 (577) | 4326 (1246) | 4909 (1022)

9. Secondary Outcome: MEDI3902 Serum Clearance (CL) of MEDI3902
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. The PK parameter CL was estimated based on the serum concentrations of MEDI3902. Non-compartmental PK data analysis was performed to estimate the serum PK parameters of MEDI3902.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milliliters/day
Arm/Group | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 3 | 15 | 15 | 8
milliliters/day | 371 (79) | 371 (101) | 373 (83) | 489 (128)

10. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) to MEDI3902
Description: Blood samples were collected to evaluate the antidrug antibody responses to MEDI3902 in serum. The number of participants positive for serum antibodies to MEDI3902 were presented.
Time Frame: Days 1 (pre-dose), 15, 29, and 61
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
Number analyzed (Participants) | 14 | 3 | 15 | 15 | 9
Participants
  Pre-dose (Baseline) | 0 | 1 | 0 | 1 | 0
  Day 15: number analyzed (Participants) | 14 | 3 | 14 | 15 | 9
  Day 15 | 0 | 0 | 0 | 0 | 0
  Day 29: number analyzed (Participants) | 14 | 2 | 15 | 14 | 9
  Day 29 | 0 | 0 | 0 | 0 | 0
  Day 61: number analyzed (Participants) | 14 | 2 | 15 | 15 | 9
  Day 61 | 1 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signature of informed consent through Day 61 of the study.
Arm/Group | Placebo | MEDI3902 - Dose 1 | MEDI3902 - Dose 2 | MEDI3902 - Dose 3 | MEDI3902 - Dose 4
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/3 | 0/15 | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/3 | 0/15 | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 4/14 | 2/3 | 6/15 | 8/15 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | MEDI3902 - Dose 1 (N=3) | MEDI3902 - Dose 2 (N=15) | MEDI3902 - Dose 3 (N=15) | MEDI3902 - Dose 4 (N=9)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 6 | 5
Headache (Nervous system disorders) | 2 | 1 | 2 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.